CLINICAL TRIAL: NCT01277107
Title: Double Blind, Polysomnographic, Two-Way Crossover Study To Compere The Efficacy Of Gastric Retentive Zaleplon (Zaleplon AP) To Placebo In Subjects With Insomnia Characterized By Both Difficulty In Falling Asleep And Staying Asleep
Brief Title: A Polysomnographic Study to Compare the Efficacy of Gastric Retentive Zaleplon Accordion Pill to Placebo in Subjects With Insomnia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Intec Pharma Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IN 09 006
Record Dates: First submitted 2011-01-12; First posted 2011-01-14 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2014-12

CONDITIONS: Insomnia
Keywords: PSG; LPS; TST; WASO; Subjects With Insomnia characterized by both Difficulty in Falling Asleep and Staying Asleep
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Zaleplon AP formulation (Experimental): Gastric Retentive Dual Release Zaleplon (Zaleplon AP)
  Interventions: Drug: Zaleplon AP formulation
- Placebo (Placebo Comparator): Identical placebo capsule
  Interventions: Drug: Placebo capsule

INTERVENTIONS:
Drug: Zaleplon AP formulation — Gastric retentive dual release Zaleplon
  Arms: Zaleplon AP formulation
Drug: Placebo capsule — Identical placebo capsule
  Arms: Placebo

SUMMARY:
This is a multi center, double blind placebo controlled, two-way crossover study in patients with Insomnia suffering from difficulty in falling asleep and staying asleep. This study intends to assess the efficacy of Zaleplon AP in improving sleep parameters, comparing to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Subjects between the ages of 18 and 65 years of age
* Subjects that meet DSM IV diagnostic criteria for Primary Insomnia
* Subjects that report a time in bed ≥6.5 and ≤9 hours
* Subjects that report on a one week sleep diary (on at least 3 of 7 nights) TST ≤6.5 hours
* Subjects that report on a one week sleep diary (on at least 3 of 7 nights)Wake time after sleep >1.0 hour
* Subjects that report on a one week sleep diary (on at least 3 of 7 nights) ≥30 minutes time to sleep onset
* On two nights of PSG screening a mean WASO of ≥60 minutes with neither night less than 45 minutes
* On two nights of PSG screening a mean LPS of ≥20 minutes with neither night less than 15 minutes
* On two nights of PSG screening a TST of ≤6.5 hours on each of the two nights
* Body mass index of 18 - 34 inclusive
* Subjects that report a median habitual bedtime between 9:00pm (21:00 hours) and 12:00am (00:00) on a one week sleep diary (based on 3 or more nights).

Exclusion Criteria:

* Participation in another drug clinical trial within 1 month prior to first screening diary day (calculated from the previous study's last dosing date).
* On screening PSG night 1 an AHI >10 (apnea hypopnea index)
* On screening PSG night 1 a PLMAI ≥10 (periodic limb movements with arousal)
* Subject has a circadian rhythm disorder including shift work or the need to travel ≥3 time zones during the course of the study
* Subject has any other sleep disorder (e.g. Restless Legs Syndrome )
* Use of any drug known to effect sleep or wake functions within 5 half lives of the drug or two weeks, whichever comes first.
* Subject with a history (past year) of alcohol or substance abuse
* Subject that needs to smoke during the sleep period time
* Subject that reports habitual napping (more than 3 times per week)
* Subject has currently or a significant history of seizures, sleep apnea or restless leg syndrome or other sleep disorders which, in the opinion of the investigator responsible, contraindicates his/her participation
* Subjects with a recent history of clinically defined GERD, peptic ulcer or any gastrointestinal surgery other than appendectomy or herniotomy which, in the opinion of the investigator responsible, contraindicates his/her participation
* Subject with any gastrointestinal disorder likely to influence drug absorption, or with any history of inflammatory bowel disease, intestinal obstruction, irritable bowel syndrome, severe gastrointestinal narrowing, or frequent nausea or emesis, regardless of etiology which, in the opinion of the investigator responsible, contraindicates his/her participation
* Subjects suffering from any Axis 1 Psychiatric Disorder that in the opinion of the investigator responsible may interfere with full participation
* Subject has significant history of cardiac, pulmonary, hepatic or renal disease or other condition or any major complication/illness which, in the opinion of the investigator responsible, contraindicates his/her participation.
* The subject has any clinically important abnormal finding as determined by a medical history, physical examination, electrocardiogram, or clinical laboratory tests, as determined by the investigator
* Subject is taking CNS-active drugs (including herbal products with CNS effects), known to affect the sleep/wake cycle including but not limited to anxiolytic, hypnotics, antidepressants, sedating H1 antihistamines, systemic steroids, anticonvulsants, narcotic analgesics, respiratory stimulants respiratory decongestants, OTC and prescription diet aids, OTC and prescription stimulants, St. John's Wort, and melatonin.
* Females who are pregnant or nursing.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2011-01; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
To determine the effect of dual release Zaleplon (Zaleplon AP) on Total Sleep Time (TST) | Polysomnography tests for 2 consecutive nights at each treatment arm
  The change from baseline on the mean of drug nights 1 and 2 relative to placebo.

SECONDARY OUTCOMES:
To determine the efficacy of Zaleplon AP on Latency to Persistent Sleep (LPS) | Polysomnography tests for 2 consecutive nights at each treatment arm
  The change from baseline on the mean of drug nights 1 and 2 relative to placebo.
To determine the efficacy of Zaleplon AP on Wake time After Sleep Onset (WASO) | Polysomnography tests for 2 consecutive nights at each treatment arm
  The change from baseline on the mean of drug nights 1 and 2 relative to placebo.
To evaluate the presence of any residual effects using the digital symbol substitution test (DSST) and a memory test | 2 consecutive mornings at each treatment arm
  The change from baseline on the mean of drug nights 1 and 2 relative to placebo.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (5):
  - Pacific Sleep Medicine, San Diego, California
  - Miami Research Associates, Miami, Florida
  - Broward Research Group, Pembroke Pines, Florida
  - CRG of St. Petersburg, St. Petersburg, Florida
  - Vince and Associates Clinical Research, Overland Park, Kansas
- Rambam sleep center, Haifa, Israel